CLINICAL TRIAL: NCT01691651
Title: Botulinum Toxin Type A for Keratoconus
Brief Title: Botulinum Toxin A for the Treatment of Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Adimara da Candelaria Renesto, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECUNIFESP-87051
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Keratoconus
Keywords: Keratoconus; Tetanus toxin
MeSH Terms: conditions — Keratoconus | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin type A (Active Comparator): The group that will be subjected to the injection of botulinum toxin (subcutaneous injection of botulinum toxin type A).Subcutaneous botulinum toxin A injection will be performed in this group, (2.5 units per point application), at two points in a nasal and temporal extent of the orbicularis muscle.
  Interventions: Procedure: Subcutaneous injection of botulinum toxin type A; Drug: Botulinum Toxin Type A
- Control (No Intervention): The group that will not be subjected to any intervention.

INTERVENTIONS:
Procedure: Subcutaneous injection of botulinum toxin type A — Subcutaneous injection of botulinum toxin type A (2.5 units per application point) at two points in a nasal and temporal extent of the orbicularis muscle will be performed in the Botulinum toxin type A group.
  Arms: Botulinum toxin type A
Drug: Botulinum Toxin Type A — 2.5 units per point of application at two points in a nasal and temporal extent of the orbicularis muscle.
  Other Names: Botox (Allergan)
  Arms: Botulinum toxin type A

SUMMARY:
The purpose of this study is to associate the use of botulinum toxin type A for patients with keratoconus to demonstrate that tension eyelid has an important role in disease progression.

DETAILED DESCRIPTION:
Subcutaneous injection of botulinum toxin type A will be performed at two points in a nasal and temporal extent of the orbicularis muscle of a group of patients with keratoconus (Botulinum toxin A group).The idea is to evaluate the change in palpebral fissure in patients from group botulinum toxin A over a period of 18 months.The measurements of the palpebral fissure will be performed by the Image J (version 1.34s) program, developed by the National Institutes of Health (USA).The unit of measure is the millimetre.The patients of the botulinum toxin A group will be compared with a control group, without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients with documented keratoconus
* best-corrected visual acuity measurable at refraction test
* age between 10-40 years
* good health
* understand the procedure and its limitations

Exclusion Criteria:

* only one functional eye
* previous ocular surgery
* concurrent corneal infection and other ocular diseases that modified the visual acuity
* known allergy to botulinum toxin
* pregnancy
* poor collaboration for performing the examinations and the procedure

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the palpebral fissure | Eighteen months.
  We will evaluate the change in palpebral fissure (unit of measure=millimetre)by 18 months.These time points will be included:baseline, 3, 6, 12 and 18 months.

SECONDARY OUTCOMES:
Corneal topography | Eighteen months.
  We will evaluate corneal topography [flattest keratometry, steepest keratometry and average keratometry(unit of measure=diopters)]by 18 months.These time points will be included:baseline, 3, 6,12 and 18 months.

OTHER OUTCOMES:
Corrected visual acuity | Eighteen months.
  We will evaluate the corrected visual acuity (unit of measure=logMAR)by 18 months.These time points will be included:baseline, 3, 6, 12 and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adimara C Renesto, MD, Principal Investigator — Federal University of São Paulo; Teissy H Osaki, MD, Study Chair — Federal University of São Paulo; Midori H Osaki, MD, Study Chair — Federal University of São Paulo; Mauro Q Campos, MD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, Department of Ophthalmology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Edwards M, McGhee CN, Dean S. The genetics of keratoconus. Clin Exp Ophthalmol. 2001 Dec;29(6):345-51. doi: 10.1046/j.1442-9071.2001.d01-16.x. PMID 11778802
- [Background] Miranda D, Sartori M, Francesconi C, Allemann N, Ferrara P, Campos M. Ferrara intrastromal corneal ring segments for severe keratoconus. J Refract Surg. 2003 Nov-Dec;19(6):645-53. doi: 10.3928/1081-597X-20031101-06. PMID 14640429
- [Background] Kymionis GD, Kontadakis GA, Kounis GA, Portaliou DM, Karavitaki AE, Magarakis M, Yoo S, Pallikaris IG. Simultaneous topography-guided PRK followed by corneal collagen cross-linking for keratoconus. J Refract Surg. 2009 Sep;25(9):S807-11. doi: 10.3928/1081597X-20090813-09. Epub 2009 Sep 11. PMID 19772256
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Renesto Ada C, Melo LA Jr, Sartori Mde F, Campos M. Sequential topical riboflavin with or without ultraviolet a radiation with delayed intracorneal ring segment insertion for keratoconus. Am J Ophthalmol. 2012 May;153(5):982-993.e3. doi: 10.1016/j.ajo.2011.10.014. Epub 2012 Jan 20. PMID 22265143
- [Background] Bawazeer AM, Hodge WG, Lorimer B. Atopy and keratoconus: a multivariate analysis. Br J Ophthalmol. 2000 Aug;84(8):834-6. doi: 10.1136/bjo.84.8.834. PMID 10906086
- [Background] Kim T, Khosla-Gupta B, Debacker C. Blepharoptosis-induced superior keratoconus. Am J Ophthalmol. 2000 Aug;130(2):232-4. doi: 10.1016/s0002-9394(00)00497-9. PMID 11004300
- [Background] Parunovic A. Floppy eyelid syndrome. Br J Ophthalmol. 1983 Apr;67(4):264-6. doi: 10.1136/bjo.67.4.264. PMID 6830745
- [Background] Brown IA. Ankyloblepharon associated with keratoconus. Br J Ophthalmol. 1967 Feb;51(2):138-9. doi: 10.1136/bjo.51.2.138. No abstract available. PMID 6018907
- [Background] Cristina Kenney M, Brown DJ. The cascade hypothesis of keratoconus. Cont Lens Anterior Eye. 2003 Sep;26(3):139-46. doi: 10.1016/S1367-0484(03)00022-5. PMID 16303509
- [Background] Scott AB, Kennedy RA, Stubbs HA. Botulinum A toxin injection as a treatment for blepharospasm. Arch Ophthalmol. 1985 Mar;103(3):347-50. doi: 10.1001/archopht.1985.01050030043017. PMID 3977705
- [Background] Schellini SA, Matai O, Igami TZ, Padovani CR, Padovani CP. [Essential blepharospasm and hemifacial spasm: characteristic of the patient, botulinum toxin A treatment and literature review]. Arq Bras Oftalmol. 2006 Jan-Feb;69(1):23-6. doi: 10.1590/s0004-27492006000100005. Epub 2006 Feb 10. Portuguese. PMID 16491229
- [Background] Nicoletti AG, Aoki L, Nahas TR, Matayoshi S. [Essential blepharospasm: literature review]. Arq Bras Oftalmol. 2010 Sep-Oct;73(5):469-73. doi: 10.1590/s0004-27492010000500018. Portuguese. PMID 21225137
- [Background] Coscarelli JM. Essential blepharospasm. Semin Ophthalmol. 2010 May;25(3):104-8. doi: 10.3109/08820538.2010.488564. PMID 20590421
- [Background] Krumeich JH, Daniel J, Knulle A. Live-epikeratophakia for keratoconus. J Cataract Refract Surg. 1998 Apr;24(4):456-63. doi: 10.1016/s0886-3350(98)80284-8. PMID 9584238
- [Derived] Renesto ADC, Osaki TH, Osaki MH, Hirai FE, Campos M. Keratoconus progression is not inhibited by reducing eyelid muscular force with botulinum toxin A treatment: a randomized trial. Arq Bras Oftalmol. 2017 Mar-Apr;80(2):88-92. doi: 10.5935/0004-2749.20170022. PMID 28591280
- See also: Pubmed comprises citations for biomedical literature from MEDLINE, life science journals, and online books. — http://pubmed.gov